CLINICAL TRIAL: NCT00769535
Title: Relationship Between Polymorphism of Heat Shock Protein 70 Gene and Hepatocellular Carcinoma
Acronym: HSP70
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KMUH-IRB-930047
Record Dates: First submitted 2008-02-26; First posted 2008-10-09 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: heat shock protein70; tumor necrosis factor-alpha promoter; polymorphism
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSP70 and TNF polymorphisms (Experimental)
  Interventions: Genetic: Polymorphisms of HSP70 and TNF promoter

INTERVENTIONS:
Genetic: Polymorphisms of HSP70 and TNF promoter — To assess the relationship between clinical relevance and polymorphisms of HSP70 and tumor necrosis factor-alpha with PCR_RFLP
  Other Names: polymorphism of HSP70; polymorphism of tumor necrosis factor-alpha promoter

SUMMARY:
Polymorphisms of HSP70 and tumor necrosis factor-alpha promoter in patients with hepatocellular carcinoma, chronic liver disease and healthy controls will be measured by PCR-RFLP or direct sequencing. The clinical relevance of patients will be compared in those with polymorphism and those without.

DETAILED DESCRIPTION:
Heat shock protein 70 (HSP 70) may be involved in various aspects of immune system including infection, autoimmunity, and tumor immunity. The relationship between HSP70 expression, disease activity and cancer prognosis varied according to type of cancer. The overexpression of HSP70 by tumor cells contributes to tumor behavior. HSP70 is present in normal and abnormal hepatocytes, and was reported to be over-expressed in both hepatoma cell lines and human hepatocellular carcinoma (HCC) tissue. Recent study indicated that HSP70 is a molecular marker during early hepatocarcinogenesis. It is also involved in anti-tumor immunity in HCC.We also investigate the polymorphism of tumor necrosis factor-alpha promoter, and correlated to clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* History proven HCC patients

Exclusion Criteria:

* No-definite diagnosed patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Clinical relevance | year

SECONDARY OUTCOMES:
Clinical relevance | year

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Fa Tsai, M.D., Ph.D., Principal Investigator — Professor of Medicine
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University, Kaohsiung City, Kaohsiung
  - Kaohsiung Medical University, Kaohsiung City, Kaohsiun